CLINICAL TRIAL: NCT02927691
Title: Novel Management of Airway Protection in Parkinson's Disease: A Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 542528
Record Dates: First submitted 2016-09-13; First posted 2016-10-07 (Estimated); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease; Dysphagia; Dystussia
Keywords: Rehabilitation; Parkinson's disease; Swallowing; Cough; Dysphagia; Dystussia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Treatment (Experimental): Participants will begin treatment immediately following baseline testing.
  Interventions: Device: EMST; Behavioral: smTAP
- Delayed Treatment (Other): Following baseline testing, participants will receive no treatment for five weeks, then begin treatment immediately following a second baseline testing session.
  Interventions: Device: EMST; Behavioral: smTAP

INTERVENTIONS:
Device: EMST
Behavioral: smTAP

SUMMARY:
Currently, there are no efficacious behavioral treatment approaches to address uncompensated aspiration, or aspiration without appropriate cough response, in Parkinson's disease (PD). This is of particular public health concern given that aspiration pneumonia is the leading cause of death in persons with PD. The overarching aim of the proposed study is to determine the efficacy of two distinct intensive rehabilitation paradigms, expiratory muscle strength training (EMST) and sensorimotor treatment for airway protection (smTAP), on airway protective clinical outcomes in persons with PD and dysphagia. The investigators anticipate the results will lead to reductions in the risks associated with airway protective deficits.

DETAILED DESCRIPTION:
Study Rationale:

Aspiration pneumonia is a leading cause of death in persons with Parkinson's disease (PD). One of the main reasons people with PD develop aspiration pneumonia is that they often have both swallowing dysfunction (dysphagia) and cough dysfunction (dystussia). Because of this, if food or liquid enters the airway, a cough is not elicited and the material remains in the airway (silent aspiration). It is then possible for the material to enter the lungs resulting in an infection called aspiration pneumonia. Currently, there are no tested treatment approaches that specifically target silent aspiration.

Hypothesis:

The goal of this study is to determine how well two different rehabilitation treatments, expiratory muscle strength training (EMST) and sensorimotor treatment for airway protection (smTAP), work to improve cough and swallowing function in persons with PD and dysphagia.

Study Design:

This study will include two participant groups; one group will receive EMST and the other will receive smTAP. There will be initial baseline testing of swallowing, coughing, respiratory, and laryngeal function. The investigators will also measure the participants' perception of their cough and swallowing problem. Then, participants will be randomly assigned (much like the flip of a coin) to either the EMST or smTAP training groups. The participants will be further randomized to receive immediate training or delayed training where there is a 5-week wait to start with a second baseline performed at the end of the 5-week delay. Once training is complete the participants will once again complete measures of swallowing, coughing, respiratory and laryngeal function.

Impact on Diagnosis/Treatment of Parkinson's Disease:

The investigators anticipate that this study will assist in better understanding what treatments work best to improve swallowing and cough in people with PD; resulting in an immediate shift in the clinical management of swallowing and cough dysfunction in PD. The investigators also believe that participants will have improvements in swallowing and cough function; therefore, reducing the risk of aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PD (Hoehn and Yahr Stages II-IV)
2. Difficulty swallowing
3. Not actively receiving swallowing therapy.

Exclusion Criteria:

1. Other neurological disorders (e.g., multiple sclerosis, stroke, etc.)
2. History of head and neck cancer
3. History of breathing disorders or diseases (e.g., COPD)
4. History of smoking in the last five years
5. Uncontrolled hypertension
6. Difficulty complying due to neuropsychological dysfunction

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-09; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Troche MS, Curtis JA, Sevitz JS, Dakin AE, Perry SE, Borders JC, Grande AA, Mou Y, Vanegas-Arroyave N, Hegland KW. Rehabilitating Cough Dysfunction in Parkinson's Disease: A Randomized Controlled Trial. Mov Disord. 2023 Feb;38(2):201-211. doi: 10.1002/mds.29268. Epub 2022 Nov 7. PMID 36345090

RESULTS

PARTICIPANT FLOW:
Groups:
- Expiratory Muscle Strength Training (EMST): Participants will receive Expiratory Muscle Strength Training. Expiratory Muscle Strength Training is a device driven strength training paradigm for respiratory muscles. Twenty-five repetitions per day (5 sets of 5 repetitions) will be completed five days per week. Once per week with a clinician.
- Sensorimotor Training for Airway Protection (smTAP): Participants will be randomized to receive Sensorimotor Training for Airway Protection. Sensorimotor Training for Airway Protection is a skill-based paradigm for improving airway protective function. Twenty-five repetitions per day (5 sets of 5 repetitions) will be completed five days per week. Once per week with a clinician.
Period: Overall Study
Arm/Group | Expiratory Muscle Strength Training (EMST) | Sensorimotor Training for Airway Protection (smTAP)
Started | 34 | 31
Completed | 30 | 28
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: 65 participants were randomly assigned to either the EMST (n = 34) or smTAP (n = 31) group. Both groups should demonstrate similar demographic characteristics, including age, duration from symptom onset, and disease severity based on randomization. All 65 participants will be analyzed with intent-to-treat statistical analyses.
Groups:
- Expiratory Muscle Strength Training (EMST): Participants will receive Expiratory Muscle Strength Training (EMST)
- Sensorimotor Training for Airway Protection (smTAP): Participants will receive Sensorimotor training for airway protection (smTAP)
- Total: Total of all reporting groups
Arm/Group | Expiratory Muscle Strength Training (EMST) | Sensorimotor Training for Airway Protection (smTAP) | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 25 | 22 | 47
Age, Continuous [Mean (Full Range); unit: years] | 70.5 [53 to 87] | 69.1 [53 to 81] | 70 [53 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65
Maximum Expiratory Pressure [Least Squares Mean (Inter-Quartile Range); unit: cm H20] | 97 [39 to 156] | 112 [10 to 206] | 102 [10 to 206]
Voluntary Cough Peak Flow [Least Squares Mean (Full Range); unit: l/s] | 2.98 [1.25 to 6.76] | 3.05 [0.95 to 5.69] | 3.04 [0.95 to 6.76]

OUTCOME MEASURES:

1. Primary Outcome: Change in Voluntary Cough Peak Flow
Description: Peak expiratory flow rate (PEFR) was measured before (baseline) and after 5 weeks of treatment with EMST and smTAP.
Time Frame: Pre to Post treatment (Pre: Baseline and Post Treatment: 5 weeks)
Measure: Least Squares Mean (Full Range); unit: l/s
Groups:
- EMST: Participants will receive EMST
- smTAP: Participants will receive smTAP
Arm/Group | EMST | smTAP
Number analyzed (Participants) | 34 | 31
l/s | 0.17 [-2.32 to 3.85] | 0.51 [-1.07 to 5.82]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from start to finish of the study. Therefore, adverse events were assessed from baseline through study completion for each participant - which was a total of (on average) 1.5 months. In other words - adverse events were assessed for all assessment visits (before and after treatment) and for all treatment sessions and the treatment period.
Description: Adverse event definitions were no different than the traditional definitions.
  There were no reported adverse events during the study duration for any participants.
Arm/Group | EMST | smTAP
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31

LIMITATIONS AND CAVEATS:
Treatment adherence to the home program was measured via patient logs, which have potential to be unreliable. Another limitation is that capsaicin is not immediately available to clinicians, which can limit translation of our findings to clinical settings. Though this study included patients with mild to severe Parkinson's disease and dysphagia, it will be necessary to study whether these findings are replicated in a larger cohort of patients with severe Parkinson's disease and dysphagia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02927691/Prot_SAP_000.pdf